CLINICAL TRIAL: NCT01575210
Title: Clinical Trial of a New Mask Vent, Designed to Reduce Noise of Mask Venting
Brief Title: Assessment of the Performance of a New Reduced Noise Mask Vent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA210212
Record Dates: First submitted 2012-03-27; First posted 2012-04-11 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnoea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A_ washing procedure 1 (Experimental): This group will apply washing technique 1.
  Interventions: Device: CPAP mask
- Group B_washing procedure 2 (Experimental): This group will apply washing technique 2.
  Interventions: Device: CPAP mask

INTERVENTIONS:
Device: CPAP mask — A new vent CPAP mask system will be used in this trial.
  Arms: Group A_ washing procedure 1
Device: CPAP mask — A new vent CPAP mask system will be used in this trial
  Arms: Group B_washing procedure 2

SUMMARY:
As continuous positive airway pressure is the treatment of choice for OSA, a mask is vital in ensuring the effectiveness of therapy delivery. The study will evaluate the performance and usability of the new mask vent. This is done by comparing the apnea-hypopnea index (AHI) of patients, who will apply 2 different washing procedures to the new mask, at the end of the study and their baseline data obtained at the beginning of the study.The study will also assess the breathing comfort as well as obtaining subjective data on the usability of the new mask vent system.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are using ResMed mask
* Subjects willing to provide written informed consent
* Subjects who have been treated for OSA > 6 months
* Subjects who can read and comprehend English
* Subjects ≥ 18 years old
* Subjects who are using a ResMed S8 or S9 device

Exclusion Criteria:

* Patients who are pregnant
* Patient on bi level treatment
* Patients being treated for OSA < 6 months
* Patients who have a pre-existing lung disease/condition that would predispose them to pneumothorax (for example: COPD; lung cancer, fibrosis of the lungs; recent (<2 years ago) case of pneumonia or lung infection; lung injury).
* Patients who are deemed unsuitable by the researcher due to the following reasons:

  * They do not comprehend English
  * They are unable to provide written informed consent
  * They are physically unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The apnoea/hypopnoea index (AHI) will be recorded and analysed. | 12 weeks
  Breathing disruption events per hour of sleep will be measured and analysed

SECONDARY OUTCOMES:
The level of comfort patients experience while using the new mask vent | 12 weeks
  Patients will complete a questionnaire regarding the noise of the new vent
Patient's and bed partner's perceptions of the mask vent | 12 weeks
  Patients partners will complete a questionnaire regarding the noise of the mask vent

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Schindhelm, PhD, Principal Investigator — ResMed/ The University of New South Wales
Locations (1):
- ResMed Centre for Healthy Sleep, Sydney, New South Wales, Australia